CLINICAL TRIAL: NCT01559155
Title: Role of Proteasomes in a Dermatological Autoimmune Disease: Bullous Pemphigoid
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/PS-02; 2012-A00180-43 (Other: RCB number)
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Pemphigoid, Bullous; Pemphigus; Lupus Erythematosus, Cutaneous
Keywords: proteasomes; proteasome concentration; disease activity; proteolytic activity; autoantibodies; proteasome autoantibody
MeSH Terms: conditions — Pemphigoid, Bullous; Pemphigus; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — All left over plasma samples will be incorporated into the biological collection at the Nîmes University Hospital.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bullous pemphigoid: Patients in this cohort are newly diagnosed (or have not started treatment) with bullous pemphigoid
- Other bullous-like auto-immune: Patients in this cohort are newly diagnosed (or have not started treatment) with pemphigus (15 patients) or cutaneous lupus (15 patients)
- Control group: Patients in this cohort are hospitalized at the Nîmes University Hospital, and have no history of autoimmune, inflammatory or neoplastic disease. Patients are matched for age and sex with patients in the bullous pemphigoid cohort.

SUMMARY:
The primary objective of this study is to describe and compare plasmatic anti-proteasome auto-antibody concentrations among three distinct groups: (1) patients suffering from bullous pemphigoide; (2) patients suffering from other dermatological auto-immune diseases; (3) an elderly control group.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

To compare the following parameters between the 3 groups:

* plasmatic proteasome concentrations
* plasmatic proteasome proteolytic activity

To explore the potential relationships between:

* plasmatic proteasome concentrations
* plasmatic proteasome proteolytic activity
* plasmatic anti-proteasome auto-antibody concentrations
* measures of disease severity for dermatological auto-immune diseases

To characterize plasmatic anti-proteasome auto-antibodies in patients suffering from bullous pemphigoide and other dermatological auto-immune diseases (other bullous auto immune diseases: pemphigus, cutaneous lupus, ...).

To characterize the expression and the activity of proteasomes in skin samples, in plasma and in circulating mononuclear cells in patients with bullous pemphigoide.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is not taking systemic treatment
* The patient has not been treated with topical steroids for more than 15 days.

For the bullous pemphigoid group:

* clinical signs: erythematous-based lesions, especially on flexion areas of the arms and legs, not afflicting mucous membranes, and without atrophic scaring
* histology: without epidermal acantholysis

For the pemphigus group:

* patient with pemphigus

For the lupus group:

* systemic lupus patients: presence of the 4 diagnostic criteria for systemic lupus erythematosus as defined by the American College of Rheumatology (amended 1997)
* or characteristics of subacute cutaneous lupus: clinical, histological and immunological (anti-SSa)
* or clinical and histological characteristics of chronic lupus

For the control group:

* hospitalized patients with no history of auto-immune, inflammatory or evolving neoplastic disease

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding

For patients with bullous pemphigoid, pemphigus or lupus:

* The patient is taking systemic treatment
* The patient has been taking topical steroids for more than 15 days.

For the controls:

* autoimmune disease
* inflammatory disease
* evolving neoplastic disease
* surgery during the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is composed of three groups: (1) 50 patients with newly diagnosed (untreated) bullous pemphigoid, (2) 50 control patients matched for age and sex with the previous group and (3) 30 patients with other dermatological auto-immune disease (15 pemphigus + 15 cutaneous lupus).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2015-06-09 (Actual); Study Completion 2015-06-09 (Actual)

PRIMARY OUTCOMES:
Plasmatic concentration of anti-proteasome autoantibodies (ng/ml) | baseline

SECONDARY OUTCOMES:
the daily number of new lesions | baseline
  For patients suffering from bullous pemphigoid or pemphigus: the daily number of new lesions for the 3 days preceding blood sampling
Presence/absence of mucosal disease | baseline
  For patients suffering from bullous pemphigoid only
Disease duration (weeks) | baseline
  For patients suffering from bullous pemphigoid or pemphigus or lupus
% surface area | baseline
  For patients suffering from bullous pemphigoid or pemphigus or lupus: % of skin area affected in relation to total area
Puritis score | baseline
  For patients suffering from bullous pemphigoid only: severity of itching on a analog scale varying from 0 to 6
concentration of anti-PB18 antibodies, measured by ELISA | baseline
  For patients suffering from bullous pemphigoid only; U/ml
Immunohistochemistry | baseline
  For the first 10 patients suffering from bullous pemphigoid included at the Nîmes University Hospital only; Skin biopsy immunohistochemistry scores for the pan-alpha, alpha6, beta1, beta2, beta1i, beta5i and rpt5 subunits (negative, weak, moderate, strong)
Tissue DNA expression | baseline
  For the first 10 patients suffering from bullous pemphigoid included at the Nîmes University Hospital only; Skin biopsy, plasma and circulating mononuclear cell DNA expression for the pan-alpha, alpha6, beta1, beta2, beta1i, beta5i and rpt5 subunits (weighted by beta-actin)
presence/absence of oral lesions | baseline
  For patients suffering from pemphigus
Presence/absence of Nikolsky's sign | baseline
  For patients with pemphigus only
Pemphigus disease area index | baseline
  For patients with Pemphigus only; score varying from 0 to 120.
Anti-desmogleine 1 and 3 antibody concentrations | baseline
  For patients with Pemphigus only; ELISA (U/ml
CLASI score for lupus | baseline
  for lupus patients only; score varying from 0 to 70
Karnofsky's score (%) | baseline
Plasma proteasome concentration | baseline
  ng/ml
% trypsin-like plasma proteasome proteolytic activity | baseline
% chymotrypsin-like plasma proteasome proteolytic activity | baseline
% caspase-like plasma proteasome proteolytic activity | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Stoebner, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France